CLINICAL TRIAL: NCT00876759
Title: Whole-Brain Radiotherapy (WBRT) vs. WBRT and Integrated Boost Using Helical Tomotherapy for Patients With Multiple Brain Metastases - a Multicentre Randomized Phase II Trial
Brief Title: Whole-Brain Radiotherapy (WBRT) Versus WBRT and Integrated Boost Using Helical Tomotherapy for Multiple Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Prof. Dr. med. Martin Stuschke, Department of Radiation Oncology, Medical Faculty, University Duisburg-essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tomo0701
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Brain Metastases
Keywords: cerebral metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WBRT (Active Comparator): standard WBRT to a total dose of 30 Gy in 10 fractions
  Interventions: Radiation: whole brain radiotherapy
- WBRT with simulatneous boost (Experimental): The experimental group will be treated with helical tomotherapy giving 3 Gy per fraction to the whole brain up to a total dose of 30 Gy in 10 fractions and raising the prescribed dose to the brain metastases to 5 Gy per fraction. The dose fall off to the normal brain should be as steep as possible around each brain metastasis. The optic chiasm and the optic nerves should not receive more than 3.5 Gy per fraction.
  Interventions: Radiation: whole brain radiotherapy with simultaneous boost

INTERVENTIONS:
Radiation: whole brain radiotherapy — WBRT in 10 fractions to a total dose of 30Gy
  Arms: WBRT
Radiation: whole brain radiotherapy with simultaneous boost — Total dose: 10 fractions: whole brain total dose: 30Gy, metastases: total dose 50Gy
  Arms: WBRT with simulatneous boost

SUMMARY:
Brain metastases occur in 20-40% of patients with primary extracerebral tumors. Despite important advances in therapy of malignant solid tumors and treatment of 1-3 brain metastases, multiple brain metastases continue to present a significant problem in attempting to prevent progression of disease and limit morbidity associated with therapy. The majority of patients who develop brain metastases have a short survival, effective palliation being transient. The median survival after diagnosis is as low as 3-6 months. However, there is some evidence that selected patients survive prolonged periods with vigorous therapeutic approach.

Specific therapeutic options are surgery, chemotherapy, conventional fractionated whole-brain radiotherapy (WBRT) and radiosurgery. Radiosurgery allows delivering of a single high dose fraction of radiation to targets of 3-3.5 cm maximum diameter. In patients with newly diagnosed brain metastases, a rapid decrease of symptoms, local tumor response rate of 73-90% and a median survival of 7-12 month have been reported.

WBRT alone is the treatment of choice for patients with multiple brain metastases, and for patients with single brain metastases not amenable to surgery or radiosurgery. Median survival after WBRT alone is 3-6 months.

WBRT and radiosurgery boost have been shown to improve survival in RPA class I patients and in patients with favorable histological status and squamous cell or non-small cell lung tumors. All randomized trials showed improved local control with the addition of radiosurgery to WBRT (Andrews, 2004).

WBRT in conjunction with radiosurgery improves local control and reduces the risk of new distant brain metastases, but most studies support that combined radiosurgery and WBRT does not improve the overall survival expect for patients without evidence of extracranial disease.

Helical Tomotherapy (HT) allows as a sole modality a new treatment option: Using HT, the advantage of applying a highly conformal boost dose to the metastases and WBRT can be combined in one treatment session. Therefore, it allows applying a high dose to multiple brain metastases in the sense of an integrated boost. The focus of this study is to investigate the efficacy and safety of WBRT with an integrated boost using this new treatment modality in comparison to the effects of conventional WBRT alone.

The principal objective of the trial is to assess the therapeutic efficacy of WBRT as compared to WBRT combined with integrated boost with HT delivered to patients with 2-10 brain metastases of solid tumors. The secondary objective is to evaluate the safety of WBRT as opposed to WBRT combined with integrated boost as delivered by HT in patients with 2-10 brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed extracranial primary malignancy other than small cell lung cancer, germ cell tumor and lymphoma. Histological confirmation may have been from the primary tumor site, from another metastatic site, or from the metastatic brain lesion(s)
* 4-10 brain metastases, which are radiologically proven by MRI scan. The size of each metastasis must be between 3 mm and 4.0 cm in the largest diameter. Contrast-enhancements on MRI which are smaller than 3 mm in diameter are not considered. The total volume of the lesions must be smaller than 35 ml and the volume of perilesional normal brain receiving more than 4 Gy per fraction must be smaller than 40 ml. An evaluation of the latter criterion is strongly recommended for total lesions volume > 20 ml prior to randomization of the patient according to figure 1. OR
* 2-3 brain metastases, which are radiologically proven by MRI scan. The size of each metastasis must be between 3 mm and 4.0 cm in the largest diameter. Contrast-enhancements on MRI which are smaller than 3 mm in diameter are not considered. The patient should not be considered as a good candidate for stereotactic radiosurgery +/- whole brain radiotherapy.
* Each lesion has a distance of its margin to the chiasma opticum or the optic nerves of > 5 mm.
* Male or female, Age 18 years or older
* Laboratory requirements: hematological status must be documented.
* Platelets >30 x 109/l. If platelets are below 30 x 109/l then correction by transfusion is indicated before entry into the study according to institutional guidelines.
* Hemoglobin > 8 g/dl. If anemia is present to the extent that the hemoglobin is less than 8 g/dl then correction by transfusion and/or erythropoietin is indicated before entry into the study according to institutional guidelines.
* Before patient registration, written informed consent must be given according to ICH/GCP and national regulations.

Exclusion Criteria:

* Lesions located in the medulla oblongata or in the brainstem.
* Leptomeningeal metastases or meningosis carcinomatosa. If meningosis carcinomatosa is suspected on MRI, the presence of tumor cells in the liquor cerebrospinalis must be excluded prior study entry.
* Chemotherapy within 1 week prior to study treatment
* Need for systemic chemotherapy to control primary disease or extracranial metastases within 3 weeks after study treatment (assessed before randomization)
* Prior treatment for brain metastases other than chemotherapy or resection of brain metastases (with 2-10 measurable lesions remaining), prior cranial radiotherapy
* Severe coagulopathy
* Medical illnesses or psychiatric impairments which would prevent completion of protocol therapy
* Female patients who are pregnant at the time of entering the study. Women must agree to a beta-HCG pregnancy test if the possibility of pregnancy is believed to exist. Women and men of child bearing potential who are admitted to the trial will be advised that the treatment received may be teratogenic and are advised to take adequate measures to prevent conception.
* Participation in other clinical trials within 4 weeks prior registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
time to morphologic progression in the brain as evidenced on MRI (RECIST criteria) | 2 years

SECONDARY OUTCOMES:
local tumor control as evidenced by MRI | 2 years
time to neurocognitive progression | 2 years
time to deterioration of functional independence | 2 years
quality of life | 2 years
overall survival, cause of death distribution | 2 years
toxicity as evidenced by CTC-criteria | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Stuschke, MD pHD, Principal Investigator — University Duisburg-Essen, Medical Faculty, Department of Radiation Oncology
Locations (5):
- Germany (5):
  - University Duisburg-Essen, Medical Faculty, department of Radiation Oncology, Essen, North Rhine-Westphalia
  - Klinik für Strahlentherapie Charite Campus Mitte, Berlin
  - Universitätsklinikum Hamburg Eppendorf, Ambulanzzentrum des UKE GmbH, Bereich Strahlentherapie,, Hamburg
  - Jürgen Debus, Heidelberg
  - Klinik und Poliklinik für Strahlentherapie und Radiologische Onkologie, Klinikum rechts der Isar, Technische Universität München, München